CLINICAL TRIAL: NCT02021721
Title: Next Generation DNA Sequencing in Patients With Idiopathic Male Infertility
Status: Terminated | Type: Observational
Why Stopped: Lack of funding
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Hamad Medical Corporation (Industry); Weill Cornell Medical College in Qatar (Other)
Responsible Party: Sponsor
Other Study IDs: 13-00058 [JIRB]; 12195/12 (Other: HMC IRB)
Record Dates: First submitted 2013-11-22; First posted 2013-12-27 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cohort: Subjects who fulfill the inclusion criteria will be pre-identified by consultation with their attending physicians and by thorough review of the literature to establish that the disease is indeed genetic and unsolved.

SUMMARY:
Hypothesis: To identify new gene mutations that can be related to patients with idiopathic male factor infertility.

Primary Objective: To detect possible genetic abnormalities in families with more than one sibling with male infertility.

Secondary Objective: To evaluate using next generation DNA sequencing in cases of infertility

DETAILED DESCRIPTION:
Infertility involves about 15% of couples who attempt to conceive and the male factor accounts for about half of the cases. Idiopathic, azoospermia, or oligozoospermia, which may be genetically based, constitute a significant number of male infertility cases.In the recent years, there is increasing recognition of the genetic abnormalities as a cause of male infertility. Genetic factors contribute up to 15 - 30% of male infertility cases. These abnormalities may be numerical chromosomal abnormality; the most common is Klinefelter syndrome, or structural e.g. Y-chomosome microdeletion, DNA mutations or mitochondrial DNA mutations. They account for 5%-10% cases of oligozoospermia, to 15%-25% cases with non-obstructive azoospermia. In azoospermia, sex chromosome abnormalities are predominant. However, autosomal structural chromosomal abnormalities are the chief genetic cause of oligozoospermia and may be balanced or unbalanced. In a substantial proportion of cases (32% of infertile men, or 1.5% of the male population), the underlying causes are unknown (idiopathic infertility). While cytogenetic studies have been successful in revealing some causes most non-obstructive azoospermic men are still idiopathic. They are believed to carry unknown autosomal mutations based on studies of familial male infertility that often involves two or more siblings.Regulation of the complex process of spermatogenesis depends on the cooperation of many genes which are expressed at various stages of differentiation, where mitotic, meiotic cell divisions, and postmeiotic development finally lead to the spermatozoa. Identification of genes playing a crucial role in spermatogenesis is mainly based on the observations of rodents, particularly the mouse model. In humans, such identification remains largely unavailable because of the difficulty in gaining access to tissue samples from a male gonad and the limited possibilities of functional verification in humans. Hence the genetic causes of male infertility have not yet been well recognized. Next-generation sequencing (NGS) is an effective tool for Mendelian gene identification. So far, more than 30 Mendelian disease genes have been identified using NGS, including recessive and dominant diseases. NGS data can also be used to discover linkage and homozygosity intervals, as well as determine copy number number of specific intervals (Becker et al. 2011, Krawitz et al. 2010). 15, 16 The two major branches of next-generation DNA sequencing are whole-exome (WE) and whole genome (WG) sequencing. While WGS is more comprehensive and useful for population genetics or for diseases in which complex non-exonic inheritance is suspected, WES remains a more powerful, cost-effective tool for detecting rare mutations within a patient population. Our use of WGS or WES will depend on the nature of the patients recruited for the study. In cases where depth of coverage requirements are high, WES would be better-suited as it allows for 4-6 exomes to be covered at such depth for the same cost of 1 genome at 30X. This would aid in sampling rarer alleles within the population and discovering novel mutations in patients that are not present in their unaffected family members. This is especially useful in cases of diseases where wide allelic heterogeneity may exist, as patients who test negative for the most common mutations may have a novel mutation that would otherwise have been undetectable by traditional methods. Multiple members of the same family may be affected by infertility with similar or different presentations of testicular failure with different histopathologies. In the presence of normal karyotyping and Y-chromosome microdeletion, we are usually left with unknown genetic abnormality. Genetic causes of male factor infertility can be broadly assumed to be a result of either de novo mutations inherited by the patient from one of his parents or from polymorphisms circulating in the population. In both cases, a search for potential genetic causes for infertility must rely on comparison of the DNA sequence of the patient with a controlled fertile member of his family.

ELIGIBILITY:
Inclusion Criteria:

* The study will include male patients diagnosed with infertility, fitting one of the following categories:
* More than one family member complaining of male infertility
* All ethnicities will be included in this study
* Family members will be invited to join the study

Exclusion Criteria:

* Patients in whim infertility is suspected to be caused by environmental factors more than genetic factors
* Patients whose cause of infertility has already been determined by other clinical testing
* Patients fulfilling the inclusion criteria but the other affected family member could not be recruited or did not approve of being included in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with be recruited from HMC infertility clinic.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2012-11; Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Next generation sequencing | 1 hour
  Use next generation sequencing to discover novel genes

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Crystal, MD, Principal Investigator — Weill Medical College of Cornell University; Haitham El Bardisi, MD, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided